CLINICAL TRIAL: NCT01315652
Title: Evaluation of the Usefulness of a Center Specialized in the Standardized Management of Rheumatoid Arthritis: The COMEDRA Trial
Brief Title: Interest of a Standardized Monitoring of Rheumatoid Arthritis: The COMEDRA Trial
Acronym: COMEDRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: 1 French Society of Rheumatology (Unknown); Roche Chugai (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P100113; P140101 (Other: AP-HP)
Record Dates: First submitted 2011-03-09; First posted 2011-03-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: 1 Rheumatoid arthritis; 2 Education; 3 Co-morbidities; 4 Nurse
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auto DAS (Experimental): "Auto-DAS"Number of patients with a modification in their treatment between baseline and 6 months visits
  Interventions: Behavioral: Auto-DAS
- Comorbidities treatment (Active Comparator)
  Interventions: Behavioral: Comorbidities treatment

INTERVENTIONS:
Behavioral: Comorbidities treatment — " Comorbidities treatment":Number of actions initiated in order to treat or prevent Rheumatoid Arthritis comorbidities during the 6 months follow-up
  Arms: Comorbidities treatment
Behavioral: Auto-DAS — "Auto-DAS"Number of patients with a modification in their treatment between baseline and 6 months visits
  Arms: Auto DAS

SUMMARY:
The two objectives of this trial are :1 To evaluate the impact of a visit with a nurse checking the preventive modalities and/or the presence of comorbidities such as infections ( e.g. vaccinations), cardiovascular-diseases (e.g. Indication to statin, antiaggregant,anti-hypertensive treatment…), cancers (e.g.mammography,…), osteoporosis (e.g. bone densitometry,..) in patients suffering from Rheumatoid Arthritis 2 To evaluate the impact of an educational program aimed at permitting rheumatoid arthritis patients to auto-evaluate their disease activity by collecting the Disease Activity Score (DAS28-ESR).

DETAILED DESCRIPTION:
Patients with a stable definite Rheumatoid Arthritis will be invited by their rheumatologists to participate at this study in 20 centers in France. After written informed consent will be obtained, the patients will be randomized in two arms:

* comorbidities
* auto-DAS The patients will be seen again in the same center six months later in order to collect the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis
* Stable (no change in therapy)
* Adult
* Able to collaborate

Exclusion criteria

* Pregnant woman
* Change of the therapy for 3 months before the inclusion
* Alcoholism, toxicomania, psychological problem, sever co morbidity which could invalid the consent or limit the protocol compliance
* No social coverage affiliate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comorbidities treatment | 6 months later
  Number of actions initiated I order to treat or prevent Rheumatoid Arthritis comorbidities
Auto-DAS: Patient education to calculate his Disease Activity Score | 6 months after
  Number of patients with a modification in their treatment between baseline and 6 months visits

SECONDARY OUTCOMES:
Frequency of comorbidities in Rheumatoid Arthritis | 6 months later
Adhesion to the current recommendations concerning the prevention of co-morbidities | 6 months later
Compliance and satisfaction of the patients concerning the DAS educational program | 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Dougados, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gossec L, Soubrier M, Foissac F, Molto A, Richette P, Beauvais C, Ruyssen-Witrand A, Perdriger A, Chary-Valckenaere I, Mouterde G, Dernis E, Euller-Ziegler L, Flipo RM, Gilson M, Guis S, Mariette X, Pouplin S, Marhadour T, Schaeverbeke T, Sordet C, Fayet F, Dougados M. Screening for and management of comorbidities after a nurse-led program: results of a 3-year longitudinal study in 769 established rheumatoid arthritis patients. RMD Open. 2019 Jun 14;5(2):e000914. doi: 10.1136/rmdopen-2019-000914. eCollection 2019. PMID 31275607
- [Background] Gossec L, Fayet F, Soubrier M, Foissac F, Molto A, Richette P, Beauvais C, Ruyssen-Witrand A, Perdriger A, Chary-Valckenaere I, Mouterde G, Dernis E, Euller-Ziegler L, Flipo RM, Gilson M, Balandraud N, Mariette X, Pouplin S, Marhadour T, Schaeverbeke T, Sordet C, Dougados M. Is self-assessment by patients of disease activity acceptable over the long term in rheumatoid arthritis? A 3-year follow-up of 771 patients. Rheumatology (Oxford). 2019 Aug 1;58(8):1498-1499. doi: 10.1093/rheumatology/kez094. No abstract available. PMID 30915463
- [Derived] Tournadre A, Pereira B, Gossec L, Soubrier M, Dougados M. Impact of comorbidities on fatigue in rheumatoid arthritis patients: Results from a nurse-led program for comorbidities management (COMEDRA). Joint Bone Spine. 2019 Jan;86(1):55-60. doi: 10.1016/j.jbspin.2018.06.010. Epub 2018 Jul 17. PMID 30025953
- [Derived] Ferreira RJO, Dougados M, Kirwan JR, Duarte C, de Wit M, Soubrier M, Fautrel B, Kvien TK, da Silva JAP, Gossec L; CoimbRA investigators, RAID investigators and COMEDRA investigators. Drivers of patient global assessment in patients with rheumatoid arthritis who are close to remission: an analysis of 1588 patients. Rheumatology (Oxford). 2017 Sep 1;56(9):1573-1578. doi: 10.1093/rheumatology/kex211. PMID 28859325
- [Derived] Dougados M, Soubrier M, Perrodeau E, Gossec L, Fayet F, Gilson M, Cerato MH, Pouplin S, Flipo RM, Chabrefy L, Mouterde G, Euller-Ziegler L, Schaeverbeke T, Fautrel B, Saraux A, Chary-Valckenaere I, Chales G, Dernis E, Richette P, Mariette X, Berenbaum F, Sibilia J, Ravaud P. Impact of a nurse-led programme on comorbidity management and impact of a patient self-assessment of disease activity on the management of rheumatoid arthritis: results of a prospective, multicentre, randomised, controlled trial (COMEDRA). Ann Rheum Dis. 2015 Sep;74(9):1725-33. doi: 10.1136/annrheumdis-2013-204733. Epub 2014 May 28. PMID 24872377